CLINICAL TRIAL: NCT00714623
Title: A Prospective Registry for the Use of CypherTM Sirolimus-Eluting Stents In Patients With Coronary Artery Disease Treated With Percutaneous Coronary Interventions at Scripps Clinic
Brief Title: The SCRIPPS DES REAL WORLD Registry
Status: Completed | Type: Observational
Sponsor: Paul S Teirstein, MD (Other)
Collaborators: Cordis US Corp. (Industry)
Responsible Party: Sponsor-Investigator, Paul S Teirstein, MD, Chief of Cardiology, Scripps Clinic
Organization: Scripps Health (Other)
Other Study IDs: 04-048
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2012-12-24 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease; Coronary Restenosis; Coronary Thrombosis
Keywords: Coronary Artery Disease; Coronary Restenosis; Coronary Thrombosis; Drug-Eluting Stents; Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis; Coronary Thrombosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Sirolimus-Eluting Bx Velocity Coronary Stent (CypherTM Sirolimus-Eluting Stent) — Indications for use: The CYPHER™ Sirolimus-eluting Coronary Stent is indicated for improving coronary luminal diameter in patients with symptomatic ischemic disease due to discrete de novo lesions of length less than or equal to 30 mm in native coronary arteries with a reference vessel diameter between 2.5 and 3.5 mm. Long-term outcome (beyond 12 months) for this permanent implant is unknown at present.
  Other Names: CYPHER™ Stent

SUMMARY:
This study is a prospective, non-randomized, open-label registry of consecutive patients with CAD treated by stent-assisted PCI using at least one CypherTM stent. Up to 1000 pts will be included in the registry. The registry is conducted for the evaluation of the impact of CypherTM Sirolimus-eluting stent implantation in the "real world" of interventional cardiology. Informed consent will be obtained from patients meeting the inclusion criteria before the initiation of any study specific procedures. Consecutive patients treated with the use of the CypherTM stent will be included in the registry. Baseline and post-procedure blood samples will be used to perform platelet function analysis using the Accumetrics Ultegra RPFA (Rapid Platelet Function Assay).

All patients will be followed from enrollment through the hospital discharge for any clinically significant event (death, myocardial infarction, TLR, TVR, major or minor bleeding). A follow-up telephone assessment of death, myocardial infarction, revascularization, and medical treatment will be conducted by experienced research personnel at 30 days, 6 months, 1 year and at least 2 years. All site reported deaths, myocardial infarctions and revascularizations will be adjudicated by an independent Clinical Events Committee for all 1000 patients enrolled in the trial. An interim analysis of the first 750 patients will be conducted and data forwarded to FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Eligible for percutaneous coronary intervention
3. Patient has at least one lesion ≥50% diameter stenosis requiring PCI with stenting
4. Reference vessel diameter 2.25-4.0 mm
5. Percutaneous intervention with use of one or more of the FDA approved CypherTM stents, planned not to exceed 108 mm of stent length.
6. Target lesion is located within a native coronary artery or bypass graft
7. De novo and restenotic lesions, including ISR, radiation failure
8. Be reliable, cooperative and willing to comply with all protocol-specified procedures and follow-up
9. Able to understand and grant informed consent

Exclusion Criteria:

1. Confirmed pregnancy at the time of index PCI
2. Has known allergies to aspirin, and to both clopidogrel (PlavixTM) and ticlopidine (TiclidTM)
3. Has known allergies or contraindication to heparin and Bivalirudin (AngiomaxTM)
4. Known allergy or sensitivity to any component of a Sirolimus-eluting stent
5. Has a significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
6. Any serious disease condition with life expectancy of less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older undergoing PCI and requiring the placement of at least one drug-eluting stent will be included to this study. For this registry, consecutive patients, that will have coronary percutaneous intervention with the CypherTM at the Green Hospital of Scripps Clinic, will be enrolled. It is estimated that up to 1000 patients will be included in the registry enrolled over a four year period. It is expected that enrollment will conclude in March 2009.
Sampling Method: Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2005-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
1 yr target vessel failure (TVF), defined as the occurrence of any of the following within 1-year after the index procedure: death from cardiac causes, Q-wave or non-Q wave MI attributable to the target vessel (TV), or revascularization of the TV. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Teirstein, MD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Green Hospital/Scripps Clinic Torrey Pines, La Jolla, California, United States